CLINICAL TRIAL: NCT05682235
Title: Therapeutic Exercise and Education in Pain Neurophysiology to Improve Pain Intensity in Women With Endometriosis. Clinical Trial.
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valladolid (Other)
Responsible Party: Principal Investigator, Rebeca Abril Coello, Doctorate Student, University of Valladolid
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Endometriosis2022
Record Dates: First submitted 2022-12-26; First posted 2023-01-12 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-01

CONDITIONS: Endometriosis
Keywords: Pain; Quality of life; Chronic pelvic pain; therapeutic exercise; pain neurophysiology; physiotherapy
MeSH Terms: conditions — Endometriosis; Pain | interventions — Exercise Therapy; salicylhydroxamic acid

STUDY DESIGN:
Intervention Model Description: Through a randomization program, participants will be assigned to the treatment group or the control group.
Who Masked: Participant, Outcomes Assessor
Masking Description: the participants will not know in which treatment group they are, and the investigator in charge of carrying out the evaluation will not know to which group the subjects he evaluates belong to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Therapeutic Exercise AND Pain Neurophysiology Education (Experimental): Therapeutic exercise:
  Therapeutic exercise is the systematic and planned execution of posture movements and physical activities to correct or prevent alterations, improve or enhance physical functioning, prevent risk factors for solid and optimize overall health status.
  Pain Neurophysiology Education:
  Education in pain neurophysiology consists in describing to the patient the neurobiology and neurophysiology of his nervous system pain to improve the processing of it and diminish the threatening meaning of pain.
  Interventions: Other: Therapeutic exercise AND pain neurophysiology education
- Sham Comparator (Sham Comparator): Talks about healthy habits
  Interventions: Other: Sham

INTERVENTIONS:
Other: Therapeutic exercise AND pain neurophysiology education — A program of therapeutic exercise and education in the neurophysiology of pain will be applied to the participants of the experimental group and talks on healthy habits to the placebo group participants.
  Arms: Therapeutic Exercise AND Pain Neurophysiology Education
Other: Sham — Talk about healthy habits
  Arms: Sham Comparator

SUMMARY:
The objective of this study will be to evaluate treatment using ET exercise and pain education in women with endometriosis to improve pain intensity.

DETAILED DESCRIPTION:
A study will be carried out whose objective is to improve the intensity of pain in women with endometriosis through a program of therapeutic exercise and education in the neurophysiology of pain. Also as secondary variables will be observed: kinesiophobia, catastrophism and impression of global improvement with treatment.

ELIGIBILITY:
Inclusion Criteria:

* Women of reproductive age between 18 and 45 years.
* Women with a medical diagnosis of endometriosis.
* Women with visual analog scale (EVA) between 4 and 10 (moderate-severe pain) during the last 3 months in the suprapubic area, abdomen or perineum both continuously and intermittently.

Exclusion Criteria:

* Women who must have surgery during the study.
* Women who have undergone abdominal or pelvic surgery or who have given birth (vaginal or cesarean) in the last 6 months.
* Women who are pregnant or planning a pregnancy.
* Women with uncorrected pacemakers or coagulopathies, severe comorbid disorder, cancer (in the last 5 years or at present), severe mental disorders, or neuropathies affecting the nerves of the pelvis or lower extremities.
* Physiotherapy treatments or treatments related to pathology or study areas 15 days prior to the beginning of the study.
* Variations in medication in the 3 months prior to the start of the study.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Woman
Enrollment: 40 (Estimated)
Dates: Start 2022-12-12 (Actual); Primary Completion 2024-10-12 (Actual); Study Completion 2025-03-12 (Estimated)

PRIMARY OUTCOMES:
Changes in pain perception assessed using a 100mm Visual Analogue Scale (VAS) | Baseline, Up to 1 month, Up to 3 months
  The scale will be administered by one of the researchers. Minimum value 0. Maximum value 100. Higher score = Higher level of pain. Lowe and lower scores mean a better result.

SECONDARY OUTCOMES:
Changes in Kinesiofobia assessed using the Tampa Scale of Kinesiofobia (TSK) | Baseline, Up to 1 month, Up to 3 months
  The scale will be administered by one of the researchers. Minimum value 11. Maximum value 44. Higher score = Higher level of kinesiophobia. Lower and lower scores mean better results.
Changes in Catastrophism assesed using the Pain Catastrophism Scale (PCS) | Baseline, Up to 1 month, Up to 3 months
  The scale will be administered by one of the researchers. Minimum value 0. Maximum value 52. Higher score = Higher level of catastrophism. Lower and lower scores mean better results.
Impression of the overall improvement obtained with the treatment ussing the Global rating of changes scale (GROC) | Up to 6 months
  The scale will be administered by one of the researchers. Minimum value -7. Maximum value 7. Higher score = Increased improvement with treatment. Lower scores = 45 / 5.000 Resultados de traducción Resultado de traducción worsening of the patient with treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Sandra Jímenez, Doctor, Study Director — University of Valladolid; Luis Ceballos Laita, Doctor, Study Director — University Valladolid
Locations (1):
- University of Valladolid, Valladolid, Spain

IPD SHARING:
Plan to Share IPD: No
The data of the participants will only be kept by the study researchers.